CLINICAL TRIAL: NCT03599739
Title: Adjuvanted Influenza Vaccination and Morbidity and Mortality in U.S. Nursing Homes: Assessment of Vaccine Selection and Outcomes for the Follow-on Study Year
Brief Title: Adjuvanted Influenza Vaccination Year 2 Follow-On Survey
Status: Completed | Type: Observational
Sponsor: Insight Therapeutics, LLC (Other)
Collaborators: Seqirus (Industry); Brown University (Other)
Responsible Party: Sponsor
Other Study IDs: INSI-201805
Record Dates: First submitted 2018-07-16; First posted 2018-07-26 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Influenza; Influenza-like Illness; Influenza, Human
Keywords: Influenza; Vaccine; Vaccination; Nursing Home; Respiratory-Related Hospitalizations
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Follow-On Cohort: We will survey 823 nursing facilities who participated in the aTIV Influenza Vaccination and Morbitiy and Mortality in U.S. Nursing Homes study in 2016-2017. We anticipate a 70% response rate from this sample for participation.
  Interventions: Biological: Influenza
- Parallel Cohort: We will survey an additional 1000 facilities (i.e., facilities not participating in the original 2016-2017 study, but meeting the same entry criteria, except prior use of high dose vaccine will be allowed) in order to capture a cohort that used a wide range of self-selected vaccine choices. We anticipate a 50% response rate from this sample.
  Interventions: Biological: Influenza

INTERVENTIONS:
Biological: Influenza — Facilities will be asked to complete a survey to evaluate the impact of the influenza vaccine choice on hospitalization risk for the 2017-2018 influenza season.

SUMMARY:
The purpose of this study is to determine if different influenza vaccines produce different outcomes in nursing facility residents receiving the required annual influenza vaccination.

DETAILED DESCRIPTION:
This study will enroll facilities who participated in the adjuvanted influenza vaccine study in 2016-2017 to document the vaccine choice for the 2017-2018 influenza season through a survey. Additional facilities will be enrolled that did not participate to answer a survey responding to questions regarding the vaccine choice for the 2017-2018 and 2018-2019 flu season. Both groups will also gather information on vaccination rates for residents and staff, policies and procedures, and influenza outbreaks.

The facility will complete a profile and answer questions regarding influenza vaccination in their facilities for the 2017-2018 and 2018-2019 flu seasons.

The study team will obtain data from the Centers for Medicare & Medicaid Services in 2019 to determine the study outcomes. None of the data used in the analysis will be linked to individual residents in facilities.

ELIGIBILITY:
Inclusion Criteria:

* Participated in the Adjuvanted Influenza Vaccination and Morbidity and Mortality in U.S. Nursing Homes study
* OR
* Long-term care facilities within 75 miles of one of the 121 cities that serve as CDC surveillance sites

Exclusion Criteria:

* Facilities having fewer than 50 long-stay residents
* Hospital based facilities
* Facilities with more than 20% of the population under age 65
* Facilities not submitting Minimum Data Set (MDS) data

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Long-term care facilities within 75 miles of one of the 121 cities that serve as CDC surveillance sites. These facilities must not have fewer than 50 long-stay residents, facilities that are hospital based, facilities with more than 20% of the population under age 65, and facilities not submitting Minimum Data Set (MDS) data.
Sampling Method: Non-Probability Sample
Enrollment: 598 (Actual)
Dates: Start 2018-07-13 (Actual); Primary Completion 2019-02-15 (Actual); Study Completion 2023-01-25 (Actual)

PRIMARY OUTCOMES:
Hospitalization for all causes | up to 1 year
  Time to first occurrence of hospitalization for all-causes.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Gravenstein, MD, MPH, Principal Investigator — Brown University; Vincent Mor, PhD, Principal Investigator — Brown University; Pedro Gozalo, Phd, Principal Investigator — Brown University; H. Edward Davidson, PharmD, MPH, Principal Investigator — Insight Therapeutics, LLC
Locations (1):
- Insight Therapeutics, LLC, Norfolk, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] DiazGranados CA, Dunning AJ, Robertson CA, Talbot HK, Landolfi V, Greenberg DP. Effect of Previous-Year Vaccination on the Efficacy, Immunogenicity, and Safety of High-Dose Inactivated Influenza Vaccine in Older Adults. Clin Infect Dis. 2016 May 1;62(9):1092-1099. doi: 10.1093/cid/ciw085. Epub 2016 Feb 21. PMID 26908801
- [Background] Flannery B, Chung JR, Thaker SN, Monto AS, Martin ET, Belongia EA, McLean HQ, Gaglani M, Murthy K, Zimmerman RK, Nowalk MP, Jackson ML, Jackson LA, Foust A, Sessions W, Berman L, Spencer S, Fry AM. Interim Estimates of 2016-17 Seasonal Influenza Vaccine Effectiveness - United States, February 2017. MMWR Morb Mortal Wkly Rep. 2017 Feb 17;66(6):167-171. doi: 10.15585/mmwr.mm6606a3. PMID 28207689
- [Background] Gravenstein S, Davidson HE, Taljaard M, Ogarek J, Gozalo P, Han L, Mor V. Comparative effectiveness of high-dose versus standard-dose influenza vaccination on numbers of US nursing home residents admitted to hospital: a cluster-randomised trial. Lancet Respir Med. 2017 Sep;5(9):738-746. doi: 10.1016/S2213-2600(17)30235-7. Epub 2017 Jul 20. PMID 28736045
- See also: Australian Influenza Surveillance Report and Activity Updates, Australian Influenza Surveillance Report No. 05 - 08 July to 21 July 2017 — http://www.health.gov.au/flureport